CLINICAL TRIAL: NCT02598102
Title: Efficacy of Preprocedural Diclofenac in Males Undergoing Double J Stent Removal Under Local Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Nephro Urology, Bangalore (Other Government)
Responsible Party: Principal Investigator, Vilvapathy Senguttuvan Karthikeyan, MCh Urology Postgraduate in Urology, Institute of Nephro Urology, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INU/RRC/01/2014-15
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac sodium (Experimental): Oral diclofenac 75 mg one hour prior to stent removal
  Interventions: Drug: Diclofenac sodium
- Placebo (Placebo Comparator): Placebo one hour prior to stent removal
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac sodium — Diclofenac for pain relief
  Other Names: Voveran
  Arms: Diclofenac sodium
Drug: Placebo — Placebo for comparison
  Arms: Placebo

SUMMARY:
Double J (DJ) stents are placed following upper urinary tract surgeries. DJ stents are usually removed under local anesthesia using rigid cystoscope. Patients experience a lot of pain during this procedure and also continue to have discomfort during voiding for few days. The use of lignocaine jelly during this procedure is not very effective. Use of diclofenac suppository during flexible cystoscopy has been proven to be effective. This study was done to assess the effect of oral diclofenac in pain relief in patients undergoing DJ stent removal by rigid cystoscopy when compared to placebo and to assess its safety in these patients

DETAILED DESCRIPTION:
Consecutive consenting male patients undergoing DJ stent removal under local anesthesia during 2014-15 were enrolled. Patients were randomized to receive 75 mg oral diclofenac or placebo 1 hour prior to procedure by double blind randomization. Intraurethral 2% lignocaine jelly (25 ml) was used in both groups. Pain during rigid cystoscopy, pain at first void and at 24 hours after cystoscopy was assessed using visual analogue scale [VAS] (0 to 100). Adverse reactions to diclofenac and episodes of acute urinary retention, if any, were assessed.

ELIGIBILITY:
Inclusion Criteria:

All consecutive consenting male patients aged more than 18 years, undergoing DJ stent removal under local anesthesia (2% Lignocaine jelly) during the study period will be included.

Exclusion Criteria:

* Patients unable to understand visual analogue pain score
* Age < 18 years
* Presence of Lower Urinary Tract Symptoms prior to surgery
* Presence of prostatitis or urethral stricture during cystoscopy
* Patients with renal failure (Serum creatinine > 1.3 mg/dl)
* Patients on concomitant nephrotoxic drugs
* Patients with history of peptic ulcer or upper gastrointestinal bleed or upper abdominal surgeries
* Loss to follow up at 24 hours following DJ stent removal

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain | Intraoperative upto 24 hours postoperative
  Pain during stent removal, first void and 24 hours after procedure

SECONDARY OUTCOMES:
Adverse reactions | 24 hours
  Adverse reactions to diclofenac sodium

CONTACTS AND LOCATIONS:
Overall Officials: VS Karthikeyan, Principal Investigator — Postgraduate in Urology
Locations (1):
- Institute of Nephro Urology, Bangalore, Karnataka, India

REFERENCES:
- [Result] Chen YT, Hsiao PJ, Wong WY, Wang CC, Yang SS, Hsieh CH. Randomized double-blind comparison of lidocaine gel and plain lubricating gel in relieving pain during flexible cystoscopy. J Endourol. 2005 Mar;19(2):163-6. doi: 10.1089/end.2005.19.163. PMID 15798411
- [Derived] Karthikeyan VS, Keshavamurthy R, Mallya A, Chikka Moga Siddaiah M, Kumar S, Chandrashekar CR. Efficacy of preprocedural diclofenac in men undergoing double J stent removal under local anesthesia: A double-blind, randomized control trial. Indian J Urol. 2017 Jan-Mar;33(1):53-57. doi: 10.4103/0970-1591.194783. PMID 28197031